CLINICAL TRIAL: NCT07227311
Title: A Phase 2, Multicenter, Open Label, Non-randomized Study to Evaluate the Efficacy and Safety of Extended Dosing of Belantamab Mafodotin in Different Combinations With Standard of Care Regimens in Participants With Relapsed-refractory Multiple Myeloma (DREAMM-15)
Brief Title: A Study to Evaluate the Efficacy and Safety of Belantamab Mafodotin in Combination With Standard of Care in Participants With Relapsed-Refractory Multiple Myeloma (RRMM)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 224317; 2025-523117-28-00 (EU CTIS Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Relapsed-Refractory Multiple Myeloma; DREAMM-15; Belantamab Mafodotin; Blenrep; Pomalidomide; Bortezomib; Carfilzomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Dexamethasone; pomalidomide; Bortezomib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Belantamab mafodotin + Pomalidomide + Dexamethasone (BPd) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dexamethasone; Drug: Pomalidomide
- Belantamab mafodotin + Bortezomib + Dexamethasone (BVd) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dexamethasone; Drug: Bortezomib
- Belantamab mafodotin + Carfilzomib + dexamethasone (BKd) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
  Other Names: Blenrep
Drug: Dexamethasone — Dexamethasone will be administered.
Drug: Pomalidomide — Pomalidomide will be administered.
  Other Names: Imnovid
  Arms: Belantamab mafodotin + Pomalidomide + Dexamethasone (BPd)
Drug: Bortezomib — Bortezomib will be administered.
  Other Names: Velcade
  Arms: Belantamab mafodotin + Bortezomib + Dexamethasone (BVd)
Drug: Carfilzomib — Carfilzomib will be administered.
  Other Names: Kyprolis
  Arms: Belantamab mafodotin + Carfilzomib + dexamethasone (BKd)

SUMMARY:
This study is for adults with multiple myeloma (a type of blood cancer) that has come back after being treated earlier or isn't responding to the current treatment.

The main goal is to find out if the study drug, belantamab mafodotin, given less often (on an extended schedule) with other cancer medicines, can still treat the cancer effectively while causing fewer side effects, especially those affecting the eyes. The study will also look at how well the treatment works overall and how safe it is when administered to the participants.

ELIGIBILITY:
Inclusion Criteria:

• Participants are eligible to be included in the study only if all of the following criteria apply:

Applicable to All Arms - BPd, BVd, BKd:

* Male or female, 18 years or older (at the time consent is obtained).
* Have a confirmed diagnosis of Multiple Myeloma (MM) as defined by the International Myeloma Working Group (IMWG) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of zero to 2.
* Have been previously treated with at least 1, but no more than 2, prior lines of MM therapy and must have documented disease progression during or after their most recent therapy.
* Must have at least 1 aspect of measurable disease, defined as one the following:

  1. Urine M-protein excretion ≥200 mg/24 h, or
  2. Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L), or
  3. Free Light Chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum free light chain ratio (<0.26 or >1.65) only if patient has no measurable urine or serum M spike.
* Patients with a history of Autologous Stem Cell Transplant (ASCT) are eligible for study participation provided the following eligibility criteria are met:

  1. ASCT was >100 days prior to the first dose of study medication,
  2. No active bacterial, viral, or fungal infection(s) present.
* All prior treatment-related toxicities (defined by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0) must be ≤Grade 1 at the time of enrollment, except for alopecia.
* Adequate organ system functions as defined by the laboratory assessments.
* Contraceptive requirements for men and women per local regulations; strict pregnancy prevention for women of childbearing potential (WOCBP), including negative pregnancy tests and use of highly effective contraception.
* Male participants must refrain from sperm donation and must use a condom plus an additional highly effective method of contraception if sexually active with a woman of childbearing potential.

Specific Inclusion Criteria for BPd arm:

• Prior treatment must include a lenalidomide-containing regimen, with lenalidomide administered for at least 2 consecutive cycles.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Applicable for all (BPd, BVd, BKd):

* Active plasma cell leukemia at Screening.
* Symptomatic amyloidosis, including active Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal plasma proliferative disorder, and Skin changes (POEMS).
* Previous or concurrent invasive malignancy other than MM, except:

  1. The disease must be considered medically stable for at least 2 years; or
  2. The patient must not be receiving active therapy, other than hormonal therapy for this disease.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Plasmapheresis within 7 days prior to the first dose of study intervention.
* Patients after prior allogeneic stem cell transplant
* Any major surgery within 4 weeks prior to start of treatment, except for bone stabilizing surgery.
* Evidence of active mucosal or internal bleeding.
* Intolerance or contraindications to anti-viral prophylaxis.
* Current corneal epithelial disease except for mild punctate keratopathy.
* Systemic anti-myeloma therapy (including chemotherapy and systemic steroids); prior treatment with an anti-MM monoclonal antibody drug within 30 days of receiving the first dose of study intervention.
* Presence of active renal condition (infection, requirement for dialysis, or any other condition that could affect participant's safety). Patients with isolated proteinuria resulting from MM are eligible, provided they fulfill certain criteria
* Received prior B-cell maturation antigen (BCMA)-targeted therapy.
* Contact lenses are prohibited while receiving belantamab mafodotin treatment. Use may be restarted after a qualified eye care specialist confirms there are no other contraindications. Bandage contact lenses are permitted during study treatment as directed by the treating eye care specialist.
* HIV infection unless well-controlled, no recent AIDS-defining infections, and adequate CD4+ count.
* Significant liver dysfunction (ALT >2.5x ULN, bilirubin >1.5x ULN, cirrhosis, unstable liver/biliary disease).
* Positive hepatitis B or C markers unless criteria for resolved infection are met.
* Evidence of cardiovascular risk including any of the following: untreated arrhythmias, recent MI/ACS/angioplasty/bypass, NYHA III/IV heart failure, uncontrolled hypertension, QTc prolongation.

Specific Exclusion Criteria for BPd Arm:

* Received prior treatment with or intolerant to pomalidomide.
* Active or history of venous and arterial thromboembolism within the past 3 months.

Specific Exclusion Criteria for BVd Arm:

* Intolerant to bortezomib or refractory to bortezomib (defined as progressive disease during treatment with a bortezomib-containing regimen of 1.3 mg/m² twice weekly or within 60 days of completing that treatment).
* Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.

Specific Exclusion Criteria for BKd Arm:

* Intolerant to carfilzomib or refractory to carfilzomib (defined as progressive disease during treatment with a carfilzomib-containing regimen or within 60 days of completing that treatment).
* Known history of allergy to captisol (i.e., cyclodextrin derivatives) used to solubilize carfilzomib.
* Left ventricular ejection fraction <40% as assessed by transthoracic echocardiogram.
* Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrolment.
* Intolerance to hydration due to pre-existing pulmonary or cardiac impairment.
* Known pulmonary hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2030-07-10 (Estimated); Study Completion 2030-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 54 months
  ORR is defined as the percentage of participants with a confirmed partial response [PR] or better (i.e., PR, very good partial response (VGPR), complete response [CR], stringent complete response [sCR]). Responses will be assessed using International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to approximately 54 months
  CRR is defined as the percentage of participants with a confirmed CR or better (i.e., CR, sCR).
Minimal Residual Disease (MRD) Negativity Rate | Up to approximately 54 months
  MRD negativity rate is defined as the percentage of participants who achieve MRD negative status (as assessed by Next generation sequencing [NGS] at 10^-5 threshold) at least once during the time of confirmed CR or better response as per IMWG.
Duration of Response (DoR) | Up to approximately 54 months
  DoR is defined as the time from first documented evidence of PR or better until PD or death due to any cause.
Number of participants with adverse events (AEs), Serious adverse events (SAEs) by severity | Up to approximately 54 months
Number of participants with AEs leading to dose modifications or AEs leading to treatment discontinuation | Up to approximately 54 months
Number of Participants With Ocular Findings on Ophthalmic Examination by severity | Up to approximately 54 months
Proportion of participants showing concordance between patient-reported ocular symptoms and ophthalmic examination findings | Up to approximately 54 months
  Ophthalmic examination findings will be summarized, and contingency table will be constructed to assess the concordance between the results from patient questionnaires (Ocular Surface Disease Index [OSDI], PRO-CTCAE ocular scale, and PROSIM-Q) and findings from clinician assessments (CTCAE for eye disorders and Keratopathy and Visual Acuity [KVA] grading scale). The proportion of participants showing concordance will be calculated from this analysis.

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf